CLINICAL TRIAL: NCT01188902
Title: The Metabolic Effect of Walnut Consumption in Healthy Men and Healthy Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Klaus Parhofer, Professor of Medicine, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Walnut-2010
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Healthy
MeSH Terms: interventions — PR-10 protein, walnut birch pollen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- walnut (Experimental): western type diet with 48 g walnut per day
  Interventions: Dietary Supplement: walnut
- control (No Intervention)

INTERVENTIONS:
Dietary Supplement: walnut — walnut consumption 48 g/d
  Arms: walnut

SUMMARY:
The objectives of the proposed study are to assess the effect of walnut consumption on parameters of lipid metabolism, glucose metabolism, incretins and adipokines, endothelial function and blood pressure in healthy men and healthy postmenopausal women

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal healthy women and healthy men
* Age > 50 yrs

Exclusion Criteria:

* Evidence of alcohol, tabacco or drug abuse
* Obesity ≥ 35 kg/m2
* Diabetes mellitus
* Hypertension
* LDL-cholesterol > 190 mg/dl, Triglycerides > 350 mg/dl
* History of atherosclerotic disease

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Fasting non-HDL-cholesterol | 8 weeks

SECONDARY OUTCOMES:
area under the triglyceride curve (AUC-TG) | 8 weeks
  area under the plasma triglyceride concentration curve following a standardized oral fat challenge
incremental area under the triglyceride curve (iAUC-TG) | 8 weeks
  incremental area under the plasma triglyceride concentration curve following a standardized oral fat challenge
LDL-cholesterol | 8 weeks
  fasting plasma LDL-cholesterol concentration
HDL-cholesterol | 8 weeks
  fasting plasma HDL-cholesterol concentration
triglyceride | 8 weeks
  fasting plasma triglyceride concentration
glucose | 8 weeks
  fasting plasma glucose concentration
HOMA | 8 weeks
insulin | 8 weeks
HbA1c | 8 weeks
area under the glucose curve (AUC-glucose) | 8 weeks
  area under the plasma glucose concentration curve following a standardized oral challenge
area under the insulin curve (AUC-insulin) | 8 weeks
  area under the plasma insulin concentration curve following a standardized oral challenge
endothelial function | 8 weeks
  Postprandial (mixed meal challenge) endothelial function (flow mediated dilatation, flow-independent dilatation)

CONTACTS AND LOCATIONS:
Locations (1):
- Med Dept. 2 Grosshadern, Munich, Germany